CLINICAL TRIAL: NCT03141671
Title: Randomized Phase II Study of Salvage XRT + ADT +/- Abiraterone Acetate and Apalutamide (ARN-509) for Rising PSA After Radical Prostatectomy With Adverse Features.(FORMULA-509 Trial)
Brief Title: Randomized Phase II Study of Salvage XRT + ADT +/- Abiraterone and Apalutamide for Rising PSA After RP (FORMULA-509)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Principal Investigator, Paul Nguyen, MD, Paul Nguyen, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-623
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; bicalutamide; abiraterone; Abiraterone Acetate; Prednisone; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GnRH + Bicalutamide (Experimental): * GnRH agonist injection monthly or every 3 months for 6 months
  * Bicalutamide by mouth once/day for 6 months
  * Salvage radiation (starting 4-10 weeks after initiation of ADT)
  Interventions: Drug: GnRH; Drug: Bicalutamide; Radiation: Salvage radiation
- GnRH+Abiraterone+Apalutamide+Prednisone (Experimental): * GnRH agonist injection monthly or every 3 months for 6 months
  * Abiraterone acetate by mouth once/day for 6 months
  * Prednisone by mouth once/day for 6 months
  * Apalutamide by mouth once/day for 6 months
  * Salvage radiation (starting 4-10 weeks after initiation of ADT)
  Interventions: Drug: GnRH; Radiation: Salvage radiation; Drug: Abiraterone; Drug: Prednisone; Drug: Apalutamide

INTERVENTIONS:
Drug: GnRH — -blocks the function of hormones including testosterone which prostate cancer uses to grow and spread
  Other Names: LHRHA
Drug: Bicalutamide — -blocks the function of hormones including testosterone which prostate cancer uses to grow and spread
  Other Names: Casodex
  Arms: GnRH + Bicalutamide
Radiation: Salvage radiation — Radiation
Drug: Abiraterone — -blocks the function of hormones including testosterone which prostate cancer uses to grow and spread
  Other Names: Zytiga
  Arms: GnRH+Abiraterone+Apalutamide+Prednisone
Drug: Prednisone — Prednisone is a corticosteroid. It prevents the release of substances in the body that cause inflammation. It also suppresses the immune system.
  Other Names: Deltasone
  Arms: GnRH+Abiraterone+Apalutamide+Prednisone
Drug: Apalutamide — -blocks the function of hormones including testosterone which prostate cancer uses to grow and spread
  Other Names: ARN-509
  Arms: GnRH+Abiraterone+Apalutamide+Prednisone

SUMMARY:
This research study is comparing two different combinations of androgen deprivation therapy (ADT) used together with radiation as a treatment for rising PSA after radical prostatectomy (prostate cancer).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that an intervention is being studied. In this study, the investigational agents are apalutamide and abiraterone acetate.

Currently, the best standard treatment for men with this type of prostate cancer includes radiation therapy combined with androgen deprivation therapy (ADT). ADT blocks the function of hormones including testosterone which prostate cancer uses to grow and spread. All participants in this study will receive the main standard form of ADT called a luteinizing hormone-releasing hormone agonist (LHRHA). Physicians often also use another drug called bicalutamide to help the LHRHA block hormone function. The investigators are testing whether using two newer anti-hormonal drugs called abiraterone acetate and apalutamide with LHRHA can improve cure rates compared to using bicalutamide plus LHRHA. These two drugs work together to suppress both testosterone and the receptor where testosterone binds thereby providing more potent hormone suppression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* PSA ≥ 0.1 after radical prostatectomy (value w/in 3 months of registration) AND at least 1 unfavorable risk factor listed below.

  * Gleason 8-10
  * PSA > 0.5
  * Pathologically positive lymph nodes
  * pT3 or pT4
  * PSA doubling time (DT) < 10 months
  * Negative margins
  * Persistent PSA after RP (PSA never dropped below 0.1 after RP)
  * Local/regional recurrence on imaging
  * Decipher "High risk" (a Medicare-reimbursed test for risk of metastases after prostatectomy)
* Candidate for salvage radiation and ADT treatment
* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately. Subject must have the ability to understand and willingness to sign the written informed consent document.
* 18 ≤ Age ≤ 95 at the time of consent
* ECOG Performance Status ≤ 2 (Appendix A)
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 3 months of registration.
* System Laboratory Value
* Hematological:

  * Platelet count (plt) ≥ 100,000/ µL
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Absolute neutrophil count (ANC) ≥ 1000 cells/µL
* Renal:

  --GFR1 ≥ 45 mL/min
* Hepatic and Other:

  * Bilirubin2 ≤ 1.5 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
  * Serum Albumin > 3.0 g/dL
  * Serum potassium ≥ 3.5 mmol/L
* Coagulation:

  * International Normalized Ratio (INR)
  * or Prothrombin Time (PT)
* Activated Partial Thromboplastin Time

  * (aPTT) ≤ 1.5 × ULN (unless on prophylactic or therapeutic dosing with low molecular weight heparin)
  * Cockcroft-Gault formula will be used to calculate creatinine clearance (see study procedure manual SPM)
  * In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin; if direct bilirubin is ≤1.5 × ULN, subject may be eligible
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential OR agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug.
* Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Ability to understand and comply with study procedures for the entire length of the study as determined by the site investigator or protocol designee
* Medications known to lower the seizure threshold (see list under prohibited meds) must be discontinued or substituted at least 4 weeks prior to study entry (Section 5.5)
* Use of CYP3A4 inhibitors or inducers and CYP2D6 substrates must be discontinued prior to study entry
* Able to swallow pills

Exclusion Criteria:

* Use of post-prostatectomy ADT for > 30 continuous days prior to registration (ADT defined as use of GnRH agonist, with or without an anti-androgen). However, patients with testosterone recovery after post-prostatectomy ADT are eligible (testosterone recovery defined as total testosterone > 190 ng/dL) regardless of how long they have been on ADT.
* Prior pelvic radiation unless additional radiation can be safely delivered according to the treating physician
* PSA > 15 ng/mL in screening
* History of any of the following:

  * Seizure or known condition that may predispose to seizure (e.g., prior stroke within 1 year of randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy)
  * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
* Current evidence of any of the following:

  * Uncontrolled hypertension
  * Gastrointestinal disorder affecting absorption
  * Active infection (e.g., human immunodeficiency virus [HIV] or viral hepatitis)
  * Any chronic medical condition requiring a dose of corticosteroid higher than 10 mg prednisone/prednisolone once daily
  * Any condition that, in the opinion of the site investigator, would preclude participation in this study
  * Moderate or severe hepatic impairment (Child Pugh Class B or C)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, psychiatric illness or social situations that would limit compliance with study requirements
* Individuals with a history of another malignancy are not eligible if:

  * the cancer is under active treatment or
  * the cancer can be seen on radiology scans or
  * if they are off cancer treatment but in the opinion of their oncologist have a high risk of relapse within 5 years
* Confirmed bone metastases on imaging

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PSA Progression Free Survival | Up to 5 years
  Time from randomization to PSA failure or death due to any cause

SECONDARY OUTCOMES:
Metastasis Free Survival on conventional imaging or pathologically (MFS) | Up to 5 years
  Time from randomization to distant metastasis, identified on conventional imaging (CT, bone scan, or MRI) or pathologically, or death due to any cause or censored at date last known alive.
Metastasis Free Survival only visible by PET Imaging (MFS-PET) | Up to 5 years
  Time from randomization to distant metastasis, visible only by PET portion of a PET-CT, or death due to any cause or censored at date last known alive.
Cause Specific Survival | Up to 5 years
  The interval from randomization to the date of last known follow-up alive or date of death from each of the following causes: prostate cancer, cardiovascular disease, other causes.
Overall Survival | Up to 5 years
  Time from randomization to death due to any cause or censored at date last known alive
Time to Testosterone Recovery | Up to 5 years
  Time from randomization to date at which testosterone level returns to a normal level, or censored at the date of last disease evaluation for those whose testosterone has not reached a normal level
Toxicity as measured by CTCAE v.4.0 | Up to 5 years
  Measure Grade 1-5 toxicities at study visits and follow-up using the CTCAE v.4.0 forms and determine attribution
Time to reinitiation of ADT | Up to 5 years
  Time from randomization to date at which ADT is restarted for disease progression. Censoring occurs at date of last disease evaluation for those who are not restarted on ADT.
Patient reported QOL | Up to 5 years
  Patient-reported Quality of Life will be measured by a fatigue questionnaire
Patient reported QOL | Up to 5 years
  Patient-reported Quality of Life will be measured by a questionnaire assessing symptoms related to prostate cancer
Patient reported QOL | Up to 5 years
  Patient-reported Quality of Life will be measured by a memory survey
Cardiovascular events consisting of myocardial infarction | Up to 5 years
  Time from randomization to date at which first cardiovascular event (myocardial infarction, stroke, deep venous thrombosis, or pulmonary embolism) occurs. Censoring occurs at date of last disease evaluation for those who did not have a cardiovascular event.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nguyen, MD, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center
Locations (8):
- United States (8):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute/Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No